CLINICAL TRIAL: NCT06225141
Title: Characterization and Recognition of Genetic Diseases by Photography
Acronym: AIDY
Status: Completed | Type: Observational
Sponsor: Imagine Institute (Other)
Responsible Party: Sponsor
Other Study IDs: AIDY
Record Dates: First submitted 2023-12-28; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Dysmorphology; Orphan Diseases
Keywords: artificial intelligence
MeSH Terms: conditions — Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients
  Interventions: Other: Clinical Data reuse
- Controls
  Interventions: Other: Clinical Data reuse

INTERVENTIONS:
Other: Clinical Data reuse — Clinical Data reuse

SUMMARY:
There are around 8,000 rare diseases and new ones are described every month in the scientific literature. They affect a limited number of patients. Nearly 80% of these diseases have a genetic origin and 30 to 40% of them are associated with dysmorphia. The latter can be suspected by evaluating the morphological characteristics of the patient. This medical skill, called dysmorphology, which allows a diagnosis to be made by evaluating the morphological characteristics of a patient, is based on experience. Diagnosis is often easy for relatively common diseases, but more difficult for rarer pathologies affecting few patients and often described in a single ethnicity and age of life.

The study aims to create a dataset specific to the application of methods from artificial intelligence. Extending the methodologies described to profile and extremity photographs will allow better recognition and description of dysmorphia.

This will allow to make diagnostic suggestions by comparison with the database. The Data Science team has already explored the notion of phenotypic similarity of patients.

Jean Feydy is a mathematician expert in image analysis and will ensure the scientific robustness of the study methods.

This project will conclude with the establishment of a diagnostic aid tool, integrating research results for doctors with a particular interest in developmental anomalies and intellectual disability.

ELIGIBILITY:
The patient inclusion criteria are:

* Patients having a medical genetics, maxillofacial surgery, or craniofacial surgery consultation as part of the management of a rare disease (in France, disease affecting less than 30,000 people) associated with dysmorphia at the level of the head or neck (area from the vertex to the clavicles): hypotelorism, hypertelorism, exophthalmos, brachycephaly, anterior plagiocephaly, micrognathia, microretrognathia, prognathia, low ear, oblique eyelid fissures above, oblique eyelid fissures below, narrow eyelid fissures , small mouth, anteverted nostrils, short nose, broad nose tip, broad nose bridge, prominent nose bridge.
* Patients with a confirmed diagnosis of one of the following pathologies: Noonan, 22q11.2 deletion, Crouzon, Kabuki, Pitt Hopkins, Mowat Wilson, Cornelia de Lange, Treacher-Collins, Goldenhar or by Silver-Russel
* Patients for whom photographs of the face and/or hands are taken as part of their treatment

The inclusion criteria for control subjects are:

* Patients having a maxillofacial surgery consultation, as part of the management of a disease other than a rare disease associated with dysmorphia in the head or neck: acute pathology (wound) or chronic (gynecomastia).
* Patients for whom photographs of the face and/or hands are taken as part of their treatment

The criteria for non-inclusion of patients are:

* Patients who have undergone facial or skull surgery before the first photo was taken.
* Person subject to a judicial safeguard measure.

The criteria for non-inclusion of control subjects are:

* Pathologies affecting facial symmetry (dental cellulitis, displaced fractures).
* Patient followed for dysmorphic syndrome or in whom dysmorphic syndrome has been suspected
* Person subject to a judicial safeguard measure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Recruitment will be carried out in the departments of medical genetics, maxillofacial surgery and plastic surgery and neurosurgery (functional craniofacial surgery unit) of the Necker Enfants Malades Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 935 (Actual)
Dates: Start 2022-01-02 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
Relationship between phenotypic characteristics and genotype in rare pathologies associated with dysmorphia | through study completion, an average of 1 year
  Relationship between phenotypic characteristics (based on photographs landmarks) of the face and hand from rare pathologies associated with dysmorphia and genotype.

SECONDARY OUTCOMES:
Creation of a database of landmark photographs taken as part of care and including all patients seen in consultation | through study completion, an average of 1 year
  Creation of a database of landmark photographs taken as part of care and including all patients seen in consultation
Training an algorithm using collected data for diagnostic purposes | through study completion, an average of 1 year
  Training an algorithm using collected data to develop a dysmorphological diagnosis aid tool which could be particularly useful in situations of uncommon diseases where the clinician has not yet acquired the necessary expertise to make a diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Necker enfants malades Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No